CLINICAL TRIAL: NCT02252692
Title: Relative Bioavailability of Enalapril Administered as Orodispersible Minitablets in Healthy Adults
Brief Title: Relative Bioavailability Study With Enalapril in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ethicare GmbH (Industry)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2014-000956-28
Record Dates: First submitted 2014-09-06; First posted 2014-09-30 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Heart Failure
Keywords: Bioavailability; pharmacokinetics; enalapril; enalaprilat
MeSH Terms: conditions — Heart Failure | interventions — Enalapril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Enalapril (Active Comparator): Renitec® 2 x 5 mg tablets administered at once, to be entirely swallowed with 240 ml water
  Interventions: Drug: Enalapril
- Enalapril ODMT (Experimental): 10 x 1mg of Enalapril ODMT, swallowed entirely with 240ml of water
  Interventions: Drug: Enalapril
- Enalapril ODMT dispersed (Experimental): 10 x 1mg of Enalapril ODMT, dispersed on tongue
  Interventions: Drug: Enalapril

INTERVENTIONS:
Drug: Enalapril — oral administration
  Other Names: Renitec

SUMMARY:
Phase I study in healthy adult male and female volunteers to compare the bioavailability of enalapril administered in orodispersible Minitablets with or without water in comparison to the standard galenic tablet formulation of enalapril. The standard pharmacokinetic parameters will be calculated from the bioanalytical results for enalapril and enalaprilat and compared in a descriptive statistical analysis.

DETAILED DESCRIPTION:
Trial design: Open label, randomized, 3-way cross-over, 3-treatments, 3-periods in 24 healthy male and female adult subjects.

Primary objectives:

1. To assess the relative bioavailability of 10 mg enalapril administered as orodispersible minitablets (ODMT) with water versus a standard enalapril tablet formulation (reference product: Renitec® 2 x 5 mg tablets) taken with water;
2. To assess the relative bioavailability of 10 mg enalapril administered as orodispersible minitablets (ODMT) dispersed in the oral cavity versus a standard enalapril tablet formulation (reference product: Renitec® 2 x 5 mg tablets) taken with water.

Secondary objectives:

1. To assess whether the PK of enalapril is affected when the orodispersible minitablet (ODMT) is entirely swallowed with water versus dispersion in the oral cavity.
2. To assess the general safety and tolerability including local tolerability and palatability of enalapril administered as orodispersible minitablet (ODMT).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects aged between 18 and 55 years, inclusive.
2. Body mass index (BMI) between 18.5 and 30 kg/m2 inclusive (BMI = weight/height2).
3. Non-smoker (not smoked for at least 3 months prior to screening).
4. Physical examinations, clinical laboratory values, vital signs and ECGs are clinically acceptable to the investigator.
5. Subjects must have signed an informed consent document indicating that they understand the purpose of, and procedures required for the study and are willing to participate in the study and comply with the study procedures and restrictions.

Exclusion Criteria:

1. History or evidence of clinically significant disorder (including psychiatric), condition or disease that, in the opinion of the investigator would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.
2. Women who are lactating/breastfeeding.
3. Women planning to become pregnant during the duration of the study.
4. Men with pregnant partners or whose partners plan to become pregnant during the study.
5. Positive pregnancy test (women) on screening or predose.
6. A baseline systolic BP ≥ 140 or < 90 mmHg and/or a baseline diastolic BP of ≥ 90 or <50 mmHg. A baseline ECG QTcB > 440 ms (males) or >450 ms (females) or heart rate >100 bpm.
7. Positive for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen, or hepatitis C antibodies at screening.
8. Known substance abuse (eg, alcohol, illicit or illegal drugs) within 1 year of dosing.
9. Positive test for drug or alcohol use at screening. If the retest during the screening period is negative, subject can be included.
10. Inability or unwillingness to refrain from alcohol consumption 24 hours prior to study visits and to limit consumption throughout the course of the study.
11. Has had major surgery, donated or lost 500 mL or more of blood within 2 months of the first study treatment or has a history of chronic anemia.
12. Receiving or has received any investigational drug (or is currently using an investigational drug or device) within 30 days or 5 half-lives (whichever is longer), prior to receiving the first study treatment.
13. Use of any over-the-counter or prescription medications within 7 days or 5 half-lives (whichever is longer), prior to receiving the first study treatment. However, if a subject has to use medication within 7 days of the first study drug administration, he/she can be included in the study the study if according to the investigator the medication is not relevant within the context of the trial. Paracetamol (up to 2 g per day) for analgesia, and hormonal birth control medication will be allowed.
14. Use of any herbal medicines (eg. St. John's wort), vitamins, and supplements consumed by the subject within 7 days prior to receiving the first study treatment. However, if a subject has used herbal medicines (eg, St. John's wort), vitamins, and supplements medication within 7 days of the first study drug administration, he/she can be included in the study if according to the investigator the medication is not relevant within the context of the trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2014-08; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
AUC 0-∞ | predose, 10 min, 20 min, 30 min, 45 min, 1 hour, 1.25 hours,1.5 hours, 2 hours, 2.5 hours, 3 hours, 3.5 hours, 4 hours, 4.5 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours, 36 hours, 48 hours post-dose
  Area under the serum concentration-time curve from time of administration to infinite time for enalaprilat

SECONDARY OUTCOMES:
Safety parameters | 0-48 hours post dose, at follow-up visit
  adverse events
Tolerability Outcome Parameter | Immediately and 10 minutes after orodispersible minitablet administration
  orodispersible minitablet palatability questionnaire
AUC 0-∞ | predose, 10 min, 20 min, 30 min, 45 min, 1 hour, 1.25 hours,1.5 hours, 2 hours, 2.5 hours, 3 hours, 3.5 hours, 4 hours, 4.5 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours, 36 hours, 48 hours post-dose
  Area under the serum-concentration time curve from time of administration extrapolated to infinite time for enalapil
AUC 0-t | predose, 10 min, 20 min, 30 min, 45 min, 1 hour, 1.25 hours,1.5 hours, 2 hours, 2.5 hours, 3 hours, 3.5 hours, 4 hours, 4.5 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours, 36 hours, 48 hours post-dose
  Area under the serum concentration-time curve from from administration to the last measurable concentration or last sampling time point (48h) for enalapril
AUC 0-t | predose, 10 min, 20 min, 30 min, 45 min, 1 hour, 1.25 hours,1.5 hours, 2 hours, 2.5 hours, 3 hours, 3.5 hours, 4 hours, 4.5 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours, 36 hours, 48 hours post-dose
  Area under the serum concentration-time curve from from administration to the last measurable concentration or last sampling time point (48h) for enalaprilat
Cmax | predose, 10 min, 20 min, 30 min, 45 min, 1 hour, 1.25 hours,1.5 hours, 2 hours, 2.5 hours, 3 hours, 3.5 hours, 4 hours, 4.5 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours, 36 hours, 48 hours post-dose
  Maximum serum concentration for enalapril
Cmax | predose, 10 min, 20 min, 30 min, 45 min, 1 hour, 1.25 hours,1.5 hours, 2 hours, 2.5 hours, 3 hours, 3.5 hours, 4 hours, 4.5 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours, 36 hours, 48 hours post-dose
  Maximum serum concentration of enalaprilat
tmax | predose, 10 min, 20 min, 30 min, 45 min, 1 hour, 1.25 hours,1.5 hours, 2 hours, 2.5 hours, 3 hours, 3.5 hours, 4 hours, 4.5 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours, 36 hours, 48 hours post-dose
  Time of maximum serum concentration of enalapril
tmax | predose, 10 min, 20 min, 30 min, 45 min, 1 hour, 1.25 hours,1.5 hours, 2 hours, 2.5 hours, 3 hours, 3.5 hours, 4 hours, 4.5 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours, 36 hours, 48 hours post-dose
  Time of maximum serum concentration for enalaprilat
Ae | 0-2, 2-4, 4-8, 8-12, 12-24, 24-36, 36-48 hours post-dose
  Amount of enalaprilat or the sum of enalapril and enalaprilat excreted in urine over the time interval 0-t

CONTACTS AND LOCATIONS:
Overall Officials: Jan De Hoon, Professor, Principal Investigator — Center of Clinical Pharmacology, University Hospital Leuven, Leuven, Belgium
Locations (1):
- Center for Clinical Pharmacology, UZ Leuven, Leuven, Belgium